CLINICAL TRIAL: NCT01235299
Title: Free Flap Microcirculatory Monitoring Correlates to Free Flap Temperature Assessment
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Kraemer002
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2010-11

CONDITIONS: Flap Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy subjects
- Subjects suffering from Diabetes mellitus
- Subjects suffering from peripheral arterial occlusive disease

SUMMARY:
In case of free flap failure, time is of utmost importance as salvage rates have been reported to be inversely related to the time interval between the onset of ischemia and its clinical recognition. Consecutively, monitoring of free flaps remains of major importance. Currently, combined Laser-Doppler and Spectrophotometry is available to determine microcirculation of free flaps in reconstructive surgery as a scientific method of reliable assessment of flap perfusion. The investigators thought to analyze the correlation of free flap skin temperature and free frap microcirculation as an accurate tool of postoperative flap monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 65 years

Exclusion Criteria:

* soft tissue inflammation or osteomyelitis, peripheral arterial occlusive disease, vasculitis, chronic kidney or liver disease, cardiac dysfunction, arterial hypotension and any type of vasoactive medication, i.e. ß-blockers, calcium channel blockers, nitroglycerin or equal.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from a soft tissue defect at any location of the body receiving free flap soft-tissue defect coverage at the Department of Plastic, Hand and Reconstructive Surgery, Medical School Hannover, Germany.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Correlation of cutaneous microcirculation to free flap temperature | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Hannover, Hanover, Germany

REFERENCES:
- [Derived] Kraemer R, Lorenzen J, Knobloch K, Papst S, Kabbani M, Koennecker S, Vogt PM. Free flap microcirculatory monitoring correlates to free flap temperature assessment. J Plast Reconstr Aesthet Surg. 2011 Oct;64(10):1353-8. doi: 10.1016/j.bjps.2011.04.030. Epub 2011 Jun 12. PMID 21664205